CLINICAL TRIAL: NCT06267560
Title: A Randomized Double-blind, Placebo-controlled, Multicenter Study to Evaluate the Efficacy, Safety and Tolerability of Pelacarsen (TQJ230) in US Black/African American & Hispanic Patient Populations With Elevated Lp(a) and Established Atherosclerotic Cardiovascular Disease
Brief Title: Lp(a) Lowering Study of Pelacarsen (TQJ230) in US Black/African American and Hispanic Participants With Elevated Lp(a) and Established ASCVD
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CTQJ230A12303
Expanded Access: NCT07000695 (Available)
Record Dates: First submitted 2024-02-12; First posted 2024-02-20 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-11

CONDITIONS: Elevated Lp(a) and Established Atherosclerotic Cardiovascular Disease
Keywords: Elevated Lp(a); Cardiovascular disease; Pelacarsen (TQJ230)
MeSH Terms: conditions — Cardiovascular Diseases | interventions — pelacarsen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Eligible participants will be randomized after the screening period or Guideline recommended SOC implementation period (if needed) in a 2:1 ratio to subcutaneous injections of pelacarsen (TQJ230) 80 mg QM or placebo QM either to be self-administered or administered by caregiver or site personnel approximately every 30 days for up to 12 months.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- TQJ230 (Experimental): TQJ230 80mg QM s.c.
  Interventions: Drug: TQJ230
- Placebo (Placebo Comparator): Matching placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TQJ230 — TQJ230 80mg QM s.c.
  Other Names: pelacarsen
  Arms: TQJ230
Drug: Placebo — matching placebo
  Arms: Placebo

SUMMARY:
Study CTQJ230A12303 is a randomized, double-blind placebo-controlled, Phase IIIb study to evaluate the efficacy, safety and tolerability of pelacarsen (TQJ230) 80 mg s.c. QM compared with placebo s.c. QM in US Black/African American and Hispanic participants with established ASCVD and elevated levels of Lp(a) who are treated for cardiovascular (CV) risk factors according to local practice/guidelines for the reduction of cardiovascular risk.

DETAILED DESCRIPTION:
CTQJ230A12303 is a randomized, double-blind, placebo-controlled, multi-center, Phase IIIb study to evaluate the efficacy ( measured by reduction of the Lp(a) levels) and safety of pelacarsen (TQJ230) 80mg s.c. QM compared to placebo in US Black/African American and US Hispanic participants, with established atherosclerotic cardiovascular disease (ASCVD) as evidenced by history of coronary heart disease, cerebrovascular disease or symptomatic peripheral artery disease (PAD) and elevated levels of Lp(a).

ELIGIBILITY:
Inclusion Criteria:

* Male and female US Black/African American and US Hispanic participants 18 to ≤ 80 years of age
* Lp(a) ≥ 125 nmol/L at the screening visit, measured at the Central laboratory
* On Standard of Care (SoC) therapy for risk factors other than Lp(a), including LDL-C (LDL-C lowering therapy dose stable for at least 30 days), elevated blood pressure and diabetes, at the randomization visit according to local practice/guidelines.
* Established ASCVD disease defined as documented:

  * Coronary heart disease (CHD) and/or
  * Cerebrovascular disease (CVD) and/or
  * Peripheral arterial disease (PAD):

Exclusion Criteria:

* Uncontrolled hypertension
* Heart failure New York Heart Association (NYHA) class IV
* History of malignancy of any organ system
* History of hemorrhagic stroke or other major bleeding
* Platelet count <140,000 per mm3
* Active liver disease or hepatic dysfunction
* Significant kidney disease
* Pregnant or nursing women

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 422 (Actual)
Dates: Start 2024-04-24 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Change in log-transformed Lp(a) concentration from baseline at week 52 | Baseline, week 52
  The primary aim of the study is to demonstrate the superiority of pelacarsen to placebo in lowering the Lp(a) level at 12 months of treatment in US Black/African American and US Hispanic participants with established ASCVD and a Lp(a) level of ≥ 125 nmo/L.

SECONDARY OUTCOMES:
Incidence proportion of study discontinuations due to TEAEs | Up to 52 weeks
  Incidence proportion of study discontinuations due to TEAEs will be provided
Incidence proportion of Treatment emergent adverse events (TEAEs) of special interest | Up to 52 weeks
  Incidence proportion of Treatment emergent adverse events (TEAEs) of special interest will be provided

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (101):
- United States (94):
  - Parkway Medical Center, Birmingham, Alabama
  - Synexus, Glendale, Arizona
  - Cardiology and Medicine Clinic PA, Little Rock, Arkansas
  - National Heart Institute, Beverly Hills, California
  - Alliance Clinical, Canoga Park, California
  - Valley Clinical Trials Inc, Covina, California
  - NICRs Research Center, Garden Grove, California
  - University of Calif Irvine Med Cntr, Irvine, California
  - Long Beach Clinical Trials, Long Beach, California
  - Angel City Research Inc, Los Angeles, California
  - Velocity Clinical Trials, Los Angeles, California
  - California Medical Research Associates Inc, Northridge, California
  - Stanford University Medical Center, Palo Alto, California
  - Acclaim Clinical Research, San Diego, California
  - Excel Medical Clinical Trials LLC, Boca Raton, Florida
  - C and A Clinical Trials, Cape Coral, Florida
  - Proactive Clinical Research, Fort Lauderdale, Florida
  - National Research Institute, Hialeah, Florida
  - Sister Life Research Inc, Hialeah, Florida
  - Zenith Clinical Research, Hollywood, Florida
  - Columbus Clinical Services LLC, Miami, Florida
  - Finlay Medical Research, Miami, Florida
  - Infinite Clinical Research, Miami, Florida
  - International Research Associates, LLC, Miami, Florida
  - Baptist Health Medical Group, Miami, Florida
  - A&A Research Group Inc, Miami, Florida
  - Clinical Site Partners LLC dba Flourish Research, Miami, Florida
  - Inpatient Research Clinical LLC, Miami Lakes, Florida
  - Eminat LLC, Miramar, Florida
  - CTMD Research, Palm Springs, Florida
  - DBC Research USA, Pembroke Pines, Florida
  - New Tampa Health, Tampa, Florida
  - James A Haley Veterans Hospital, Tampa, Florida
  - Cardiology Partners Clinical Research Institute, Wellington, Florida
  - Grady Health System, Atlanta, Georgia
  - Morehouse School Of Medicine, Atlanta, Georgia
  - Comprehensive Neurosciences Inc, Atlanta, Georgia
  - Atlanta Heart Specialists LLC, Tucker, Georgia
  - Synexus Clinical Research US Inc, Chicago, Illinois
  - Chicago Clinical Research Inst, Chicago, Illinois
  - Flourish Research, Grandwood Park, Illinois
  - Cardiovascular Associates Research, Covington, Louisiana
  - Omega Clinical Research, Metairie, Louisiana
  - CV Ins of the South, Opelousas, Louisiana
  - Monroe Research Llc, West Monroe, Louisiana
  - Southern Clin Research Clinic, Zachary, Louisiana
  - Sinai Ct for Throm Res and Drug Dev, Baltimore, Maryland
  - Ascension Saint Agnes Heart Care, Baltimore, Maryland
  - Johns Hopkins Univ School of Med, Baltimore, Maryland
  - Metropolitan Cardiovascular Consultants Llc, Beltsville, Maryland
  - Johns Hopkins University, Columbia, Maryland
  - Anderson Medical Research, Ft. Washington, Maryland
  - Capitol Cardiology Associates, Lanham, Maryland
  - MD Medical Research, Oxon Hill, Maryland
  - Henry Ford Hospital, Detroit, Michigan
  - Aa Mrc Mhs, Flint, Michigan
  - Aa Mrc Llc, Flint, Michigan
  - Elite Clinical Research LLC, Jackson, Mississippi
  - Stern Cardiovascular Foundation Inc, Southaven, Mississippi
  - Las Vegas Endocrinology, Henderson, Nevada
  - AB Clinical Trials, Las Vegas, Nevada
  - Clinical Research of South Nevada, Las Vegas, Nevada
  - Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - Overlook Medical Center, Summit, New Jersey
  - Jamaica Hospital Medical Center, Jamaica, New York
  - Monroe Biomedical Research, Monroe, North Carolina
  - Alliance Medical Ministry, Raleigh, North Carolina
  - Velocity Clin Research Springdale, Cincinnati, Ohio
  - Hometown Urgent Care and Research, Columbus, Ohio
  - NexGen Research, Lima, Ohio
  - Care Access Research, Easton, Pennsylvania
  - TCV Clinical Studies, Linwood, Pennsylvania
  - The Stern Cardiovascular Foundation, Germantown, Tennessee
  - Apex Cardiology Research Associates of Jackson, Jackson, Tennessee
  - Plano Primary Care Clinic, Allen, Texas
  - Pharma Tex Research, Amarillo, Texas
  - North Hills Medical Research Inc, Bedford, Texas
  - SW Family Medicine Associates, Dallas, Texas
  - David Turbay MD PLLC, El Paso, Texas
  - Ctr for Clin Rsch and Innovatn, Houston, Texas
  - Angiocardiac Care of Texas PA, Houston, Texas
  - Dallas Heart and Vascular Consultants PA, Houston, Texas
  - Epic Clinical Research, Lewisville, Texas
  - The Heart Institute of East Texas, Lufkin, Texas
  - Discovery Clinical Trials, Pflugerville, Texas
  - University of Texas Health Science Ctr, San Antonio, Texas
  - Clinical Trials of Texas, San Antonio, Texas
  - Sugar Lakes Family Practice, Sugar Land, Texas
  - Javara Research, Alexandria, Virginia
  - Virginia Heart, Falls Church, Virginia
  - Heart Care Associates P C, Hopewell, Virginia
  - Dominion Medical Associates, Richmond, Virginia
  - Virginia Commonwealth University, Richmond, Virginia
  - University of Washington, Seattle, Washington
- Puerto Rico (7):
  - Advanced Clinical Research LLC, Bayamón
  - Dr Yolanda Figueroa Private Pr, Humacao
  - CAIMED Center, Ponce
  - Research and Cardiovascular Corp, Ponce
  - Latin Clinical Trial Center Inc, San Juan
  - VA Caribbean Healthcare System, San Juan
  - Advanced Medical Research Center, San Juan

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com